CLINICAL TRIAL: NCT04207814
Title: Determinants of Repeated Spontaneous Miscarriages and Unexplained Fetal Deaths (DEFI-2)
Brief Title: Determinants of Repeated Spontaneous Miscarriages and Unexplained Fetal Deaths
Acronym: DEFI-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DEFI-2 (29BRC19.0241)
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Repeated Spontaneous Miscarriages; Fetal Deaths in Utero

STUDY DESIGN:
Intervention Model Description: Case couples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cases (Experimental)
  Interventions: Biological: biological sample

INTERVENTIONS:
Biological: biological sample — biological samples will be taken from the subjects included

SUMMARY:
The DEFI-1 study recruited 625 women witnesses and 299 of their spouses. With regard to case couples, 271 cases were recruited from the spontaneous repeated miscarriages (SRM) subgroup (≥3 spontaneous miscarriage (SM) from trimester 1 of pregnancy) and 93 from the unexplained fetal death in utero (FDIU) subgroup from trimesters 2 and 3 of pregnancy.

The main objective of the DEFI 2 study is to increase the number of case-pairs in these 2 particular subgroups to replicate the results of the genetic determinants highlighted from cases and controls with extreme phenotypes and obtain a sufficient number of women with FDIUs to identify specific determinants.

DETAILED DESCRIPTION:
The spontaneous repeated miscarriages (SRM) affect one to two fertile couples on 100, a fetal death in utero (FDIU) complicates the evolution of a pregnancy on 200. The SRM remain unexplained in 50% of the cases although a beam indirect arguments sometimes encourage to evoke a prothrombotic process and / or endothelial dysfunction, immunological disorders, an alteration of the ovarian reserve, and possibly the impact of genetic determinants. Regarding SRM, in the absence of a fetal, funicular cause or obvious preeclampsia, very diverse mechanisms are evoked depending on the placental histology (vasculoplacental, inflammatory, intervillitis, immunological, etc.). Thus, while these mechanisms remain for some to be demonstrated and are probably not unequivocal, clinicians are faced with a pressing request for therapeutic intervention on the part of patients. This is why, after having studied in DEFI-1 the 2 main constitutional thrombophilia in the 2 members of the couple, the procoagulant circulating microparticles and the generation of thrombin in the mother on the one hand, the modalities of inactivation of an X in the mother, on the other hand, a further investigation in subgroups of particular cases would be appropriate.

ELIGIBILITY:
Inclusion Criteria:

* couples whose wife is over 18 and under 40 inclusive,
* couples having undergone at least 3 unexplained SM in the first trimester or an FDIU in the trimesters 2 and 3 of pregnancy (excluding funicular and fetal causes and proven preeclampsia)
* the man must be over 18 years old.
* each member of the couple must consent to the investigation.
* Subjects benefiting from a social security scheme.

Exclusion Criteria:

* couples where the woman is under 18 or over 40,
* couples whose man is under 18,
* identified cause of SRM or FDIU
* Inability to consent for one of the members of the couple,
* refusal to participate for one of the members of the couple.
* treatment with anticoagulants or anti-aggregating platelet for women.
* Person under legal protection
* Subjects not benefiting from a social security scheme
* Refusal to participate

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2057-10-05 (Estimated); Study Completion 2057-10-05 (Estimated)

PRIMARY OUTCOMES:
Frequency difference of the determinant between the cases and the controls | 34 years
  The frequency difference of the determinant under study between the cases (studies DEFI-1 and DEFI-2) and the controls (study DEFI-1) will be measured.

SECONDARY OUTCOMES:
Occurrence of a new medical event | 34 years
  Occurrence of a new medical event in prospective follow-up will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Pasquier, MD, Study Director — Brest University Hospital in France
Locations (1):
- BREST, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.